CLINICAL TRIAL: NCT03298958
Title: Secondary Prevention Trial of Rapamycin in Patients With Resected Non-muscle Invasive Bladder Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No funding was received, no subjects were enrolled
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20170277H
Record Dates: First submitted 2017-09-26; First posted 2017-10-02 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: When it is determined that you are eligible for the study, you will be assigned by chance (like flipping a coin) to one of 2 study groups.
  * Sirolimus 0.5 mg/day for 2 years or until disease recurrence
  * Placebo
Who Masked: Participant, Investigator
Masking Description: Double-blinded for study staff (investigator) and patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Oral Tablet (Placebo Comparator): Subject will be randomized to take the Placebo once daily for 2 years or until disease recurrence
  Interventions: Drug: Placebo Oral Tablet
- Sirolimus (Rapamycin) 0.5 mg/day for 2 years (Active Comparator): Subject will be randomized to take Sirolimus (Rapamycin) 0.5mg once daily for 2 years or until disease recurrence
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Subject will be randomized to one of the 2 arms
  Other Names: Sirolimus
  Arms: Sirolimus (Rapamycin) 0.5 mg/day for 2 years
Drug: Placebo Oral Tablet — Subject will be randomized to one of the 2 arms
  Arms: Placebo Oral Tablet

SUMMARY:
The study is a multi-site Phase 3 double-blinded randomized placebo-controlled trial. Subjects are randomly assigned to receive either a placebo or oral Sirolimus: 0.5 mg daily. All subjects will be treated for 2 years or until disease recurrence. Patients will undergo endoscopic evaluation of the bladder every 3 months for the first 2 years following enrollment and then every 6 months for an additional 2 years on study. Selection of BCG immune therapy is at the discretion of the treating urologist but in general is reserved for high-risk patients. Patients concurrently receiving BCG immune therapy will receive standard BCG therapy including induction (weekly for 6 weeks) and maintenance (weekly for 3 weeks at 3 months, 6 months, and then every 6 months following tumor resection).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically) proven diagnosis of non-muscle invasive (Ta, Tis or T1) bladder cancer within 60 days prior to enrollment
* Be able to give informed consent
* Be age 18 or older
* Not be in an immunosuppressed state (e.g. HIV, use of chronic steroids)
* Not have active, uncontrolled infections
* Not be on agents known to alter rapamycin metabolism significantly
* Not have a reported history of liver disease (e.g. cirrhosis)
* Not have a prior history of non-bladder cancer unless the cancer is clinically stable and not requiring active treatment except basal cell carcinoma or squamous cell carcinoma of the skin.
* Not pregnant, or taking effective contraception before rapamycin therapy, during therapy and for 12 weeks after discontinuation of therapy.

Exclusion Criteria:

* Have muscle-invasive (≥T2) bladder cancer
* Unable to give informed consent
* Age < 18
* Immunosuppressed state (e.g. HIV, use of chronic steroids)
* Active, uncontrolled infections
* On agents known to alter rapamycin metabolism significantly
* Another cancer requiring active treatment (except basal cell carcinoma or squamous cell carcinoma of the skin)
* Patients at risk of pregnancy who are unwilling or unable to take effective contraception before rapamycin therapy, during therapy, and for 12 weeks after discontinuation of therapy.
* Individuals with a reported history of liver disease (e.g. cirrhosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Test the hypothesis that rapamycin 0.5 mg daily increases recurrence-free survival for patients with non-muscle invasive bladder cancer | Patients are treated for 2 years or until disease relapse
  Recurrence is defined as histologically-proven bladder cancer (stage CIS, Ta, T1 or ≥T2)

SECONDARY OUTCOMES:
To determine effects of rapamycin on recurrence-free survival (RFS) for subgroup of patients with non-muscle invasive bladder cancer concurrently receiving BCG immune therapy. | Patients are treated for 2 years or until disease relapse
  Recurrence is defined as histologically-proven bladder cancer (stage CIS, Ta, T1 or ≥T2)
To compare the effects of rapamycin on BCG-specific immunity during treatment of non-muscle invasive bladder cancer with maintenance BCG. | baseline and 6 months after registration
  BCG antigen-specific IFN-gamma ELISPOT responses will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No